CLINICAL TRIAL: NCT02134184
Title: The Influence of Chronic Cytomegalovirus Infection on Influenza Vaccine Responses
Brief Title: The Influence of Chronic CMV Infection on Influenza Vaccine Responses
Acronym: SLVP025
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Philip Grant, Assistant Professor of Medicine (Infectious Diseases), Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: SU-25199; 1U19AI090019-01 (NIH)
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Results first posted 2016-12-26 (Estimated); Last update posted 2023-04-19 (Actual); Status verified 2023-04

CONDITIONS: Cytomegalovirus Infections; Influenza
MeSH Terms: conditions — Cytomegalovirus Infections; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- CMV negative group (Experimental): Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  Interventions: Biological: Fluzone® 2012-2013 Formula NDC No 498281-012-50
- CMV positive group (Experimental): Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  Interventions: Biological: Fluzone® 2012-2013 Formula NDC No 498281-012-50
- Recent CMV Converters (Experimental): Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  Interventions: Biological: Fluzone® 2012-2013 Formula NDC No 498281-012-50

INTERVENTIONS:
Biological: Fluzone® 2012-2013 Formula NDC No 498281-012-50 — This vaccine is given intramuscularly
  Other Names: Trivalent inactivated influenza vaccine (TIV)

SUMMARY:
In this study we are trying to understand whether previous infection with a particular virus, namely cytomegalovirus (CMV), influences the ability of the immune system to respond to new infections or vaccinations with age.

DETAILED DESCRIPTION:
The investigators want to compare the T- and B-cell response to conventional intramuscular trivalent influenza vaccine (TIV) in elderly individuals dependent on the presence and duration of CMV infection by analyses of vaccine-induced plasmablasts, antibodies and antigen-specific T cells. Healthy volunteers, > 60 years of age, will be identified by the Stanford Blood Center based on their history of positive or negative CMV serologies. Baseline blood samples will be drawn from all study participants prior to immunization. All participants will receive a single dose of 2012-2013 licensed TIV. Volunteers will complete 3 study visits at Day 0, Day 7 and Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy, ambulatory adult 60 years of age or above.
* Self-identified by a participant after notification by Stanford Blood Center (SBC) of their group assignment based review of SBC CMV data:

  * CMV-negative: Donor has donated at least twice during the last 3 years AND donor's most recent two donations tested CMV antibody negative.
  * CMV positive longstanding infection: Donor has donated at least once within the "recent" timeframe (past three years) AND donor's most recent donation tested CMV antibody positive AND donor had at least one donation prior to 2000 that tested CMV antibody positive.
  * Recent CMV converters: Donor has donated at least once within the "recent" timeframe (past three years) AND donor's most recent two donations tested CMV antibody positive AND donor had at least two CMV negative donations in the past.
* Willing to complete the informed consent process.
* Availability for follow-up for the planned duration of the study at least 28 days after immunization.
* Acceptable medical history by review of inclusion/exclusion criteria and vital signs.

Exclusion Criteria:

* Prior off-study vaccination with the current 2012-2013 seasonal influenza vaccine
* Allergy to egg or egg products, or to vaccine components or thimerosal (TIV multidose vials only)
* Life-threatening reactions to previous influenza vaccinations.
* Active systemic or serious concurrent illness, including febrile illness on the day of vaccination
* Weight less than 110 lbs
* History of immunodeficiency (including HIV infection)
* Known or suspected impairment of immunologic function, including, but not limited to, clinically significant liver disease, diabetes mellitus treated with insulin, moderate to severe renal disease, or any other chronic disorder which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* Blood pressure >150 systolic or >95 diastolic at first study visit
* Hospitalization in the past year for congestive heart failure or emphysema.
* History of chronic Hepatitis B or C.
* Recent or current use of immunosuppressive medication, including systemic glucocorticoids (corticosteroid nasal sprays and topical steroids are permissible in all groups)
* Malignancy, other than squamous cell or basal cell skin cancer (includes solid tumors such as breast cancer or prostate cancer with recurrence in the past year, and any hematologic cancer such as leukemia).
* Autoimmune disease (including rheumatoid arthritis treated with immunosuppressive medication such as Plaquenil, methotrexate, prednisone, Enbrel) which, in the opinion of the investigator, might jeopardize volunteer safety or compliance with the protocol.
* History of blood dyscrasias, renal disease, or hemoglobinopathies requiring regular medical follow up or hospitalization during the preceding year
* Use of any anti-coagulation medication such as Coumadin or Lovenox, or anti-platelet agents such as aspirin (except up to 325 mg aspirin per day), Plavix, or Aggrenox must be reviewed by investigator to determine if this would affect the volunteer's safety.
* Receipt of blood or blood products within the past 6 months or planned receipt of blood products prior to completion of study visits.
* Medical or psychiatric condition or occupational responsibilities that preclude participant compliance with the protocol
* Inactivated vaccine 14 days prior to vaccination or planned non-study vaccination prior to completion of Visit 03 (~Day 28 after the study vaccination)
* Live, attenuated vaccine within 60 days of vaccination or planned non-study vaccination prior to completion of Visit 03 (~Day 28 after the study vaccination)
* Need an allergy immunization (that cannot be postponed) during the study period V01 to V03 (~Day 28)
* History of Guillain-Barré Syndrome
* Use of investigational agents within 30 days prior to enrollment or planned use of investigational agents prior to completion of study visits
* Donation of the equivalent of a unit of whole blood within 6 weeks or a unit of platelets within 2 weeks prior to enrollment or planned blood donation prior to completion of study visits.
* Any condition which, in the opinion of the investigator, might interfere with volunteer safety, study objectives or the ability of the participant to understand or comply with the study protocol.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cornelia L Dekker, MD, Principal Investigator — Stanford University; Jorg J Goronzy, MD, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The NIH Human Immunology Project Consortium (HIPC) data repositories (ImmPORT) may store the results of the research assays results. Genetic data that is developed in this study may be made available to other researchers through the National Center for Biotechnology Information (NCBI) databases. Results from research assays will be labeled with a unique ID code and the volunteer identity (except for age) will not be disclosed.

RESULTS

PARTICIPANT FLOW:
Groups:
- CMV Negative Group; CMV Positive Group: Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  This vaccine is given intramuscularly
- Recent CMV Converters: Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  This vaccine is given intramuscularly Recent CMV Conversion is defined as: Donor has donated at least once within the "recent" timeframe (past three years) AND donor's most recent two donations tested CMV antibody positive AND donor had at least two CMV negative donations in the past
Period: Overall Study
Arm/Group | CMV Negative Group | CMV Positive Group | Recent CMV Converters
Started | 33 | 37 | 8
Completed | 33 | 37 | 8
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- CMV Negative Group; CMV Positive Group; Recent CMV Converters: Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  Fluzone® 2012-2013 Formula: This vaccine is given intramuscularly
- Total: Total of all reporting groups
Arm/Group | CMV Negative Group | CMV Positive Group | Recent CMV Converters | Total
Number analyzed (Participants) | 33 | 37 | 8 | 78
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 16 | 1 | 29
  >=65 years | 21 | 21 | 7 | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.96 (4.52) | 67.46 (5.26) | 66.75 (3.53) | 67.21 (4.80)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 20 | 7 | 37
  Male | 23 | 17 | 1 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 33 | 36 | 8 | 77
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 31 | 36 | 8 | 75
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 33 | 37 | 8 | 78

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants From Each Arm Who Received Influenza Vaccine
Time Frame: Day 0 to Day 28
Measure: Count of Participants; unit: Participants
Groups:
- Recent CMV Converters: Participants will receive Fluzone® 2012-2013 Formula NDC No 498281-012-50
  This vaccine is given intramuscularly
Arm/Group | CMV Negative Group | CMV Positive Group | Recent CMV Converters
Number analyzed (Participants) | 33 | 37 | 8
Participants | 33 | 37 | 8

2. Secondary Outcome: Number of Participants With Related Adverse Events
Time Frame: Day 0 to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | CMV Negative Group | CMV Positive Group | Recent CMV Converters
Number analyzed (Participants) | 33 | 37 | 8
Participants | 0 | 0 | 0

3. Other Pre Specified Outcome: To Compare the T- and B-cell Response to Licensed IM TIV in Elderly Individuals Dependent on the Presence and Duration of CMV Infection by Analyses of Vaccine-induced Plasmablasts, Antibodies and Antigen-specific T Cells
Time Frame: Day 0 to Day 28
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Day 0 to Day 28 of study participation
Description: Clinical Assessment performed at each visit
Arm/Group | CMV Negative Group | CMV Positive Group | Recent CMV Converters
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37 | 0/8
Other Adverse Events (participants affected / at risk) | 1/33 | 0/37 | 0/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CMV Negative Group (N=33) | CMV Positive Group (N=37) | Recent CMV Converters (N=8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — Community Acquired Pneumonia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No